CLINICAL TRIAL: NCT00616668
Title: Early Postoperative Fitting of the Air- Limb Prosthesis for Transtibial Amputees
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-07-2718-AK-CTIL
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Vascular Diseases
Keywords: Transtibial amputees due to vascular diseases.
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Air- Limb

SUMMARY:
The aim of the study is to check whether an early adjustment of the Air-Limb prosthesis to Transtibial amputees due to vascular diseases, will shorten the healing time of the stump and the process of rehabilitation.

DETAILED DESCRIPTION:
The method of immediate adjustment of a temporary Prosthesis has been developed in the past, aiming to reduce the healing time of the stump and the process of rehabilitation. According to this method, a temporary Prosthesis is being adjusted immediately after amputation, or during the first week after it. Rehabilitation starts with the patient's standing while partial weight bearing on the Prosthesis.

In spite of many experiments and trials to adopt this process of rehabilitation, it is not universally adopted, because of the bad adjustment and damages to the stump caused by the Plaster of Paris. At present, with the improvement of materials and research experiments are being renewed, to check the efficiency of the process, using the Air- Limb a temporary Prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Transtibial amputees due to vascular diseases.

Exclusion Criteria:

* Bilateral amputation.
* Upper extremity can't bear weight.
* The sound leg can't bear weight.
* Amputee that needs Dialysis treatment.
* Cognitive impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-01; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The duration of rehabilitation of transtibial amputees, from amputation until the fitting of the permanent prosthesis. | 1-4 month
The total duration of the rehabilitation process,from amputation until the end of the hospitalization, with the permanent prosthesis. | 2-6 month

SECONDARY OUTCOMES:
The duration of stump healing and functional status of transtibial amputees. | 1-6 month

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Siev- Ner, MD, Study Director — Sheba Medical Center